CLINICAL TRIAL: NCT06886646
Title: SCARR: Allogeneic Umbilical Cord Mesenchymal Stromal Cells for the Treatment of Chronic Antibody-Mediated Rejection (cABMR) in Kidney Transplantation
Brief Title: Allogeneic Umbilical Cord Mesenchymal Stromal Cells for the Treatment of Chronic Antibody-Mediated Rejection in Kidney Transplantation
Acronym: SCARR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: APHP220666; 2023-506598-36-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-04; First posted 2025-03-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chronic Antibody-mediated Rejection (cABMR)
Keywords: Kidney transplantation; Mesenchymal Stromal Cells (MSCs); Umbilical cord-derived MSCs
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Multicenter, controlled, randomized, double-blind, two-parallel-arm Phase II trial b. The study will be offered to eligible patients during a routine consultation. After informed consent, patients will be randomly assigned to either the CSM group or the control group (placebo (0.9% NaCl). Immunosuppressive treatment will remain unchanged in both groups.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (CSM Group) (Experimental): Patients in this arm will receive 4 injections of allogeneic mesenchymal stromal cells (CSM) derived from human umbilical cord. The doses will be 1.106 cells/kg administered intravenously at days 0, 7, 14, and 21. The injections are given after thawing, washing, resuspension, and adjusting the dose. The CSM treatment aims to control chronic active antibody-mediated rejection (cABMR), improve renal function, reduce proteinuria, and increase graft survival without changing the immunosuppressive regimen.
  Interventions: Other: Allogeneic Mesenchymal Stromal Cell Therapy
- Arm 2 (Control Group) (Placebo Comparator): Patients in this arm will receive placebo treatments, which will consist of 150 mL of saline (NaCl 0.9%) administered intravenously at the same intervals as the CSM group (days 0, 7, 14, and 21). The placebo will be administered under the same conditions as the treatment, and the participants and investigators will remain blinded to the group allocation. Like the CSM group, no changes will be made to the patients' immunosuppressive regimen.
  Interventions: Other: Placebo (NaCl 0.9%) Treatment

INTERVENTIONS:
Other: Allogeneic Mesenchymal Stromal Cell Therapy — Patients in this arm will receive 4 injections of allogeneic mesenchymal stromal cells (CSM) derived from human umbilical cord. The doses will be 1.106 cells/kg administered intravenously at days 0, 7, 14, and 21. The injections are given after thawing, washing, resuspension, and adjusting the dose. The CSM treatment aims to control chronic active antibody-mediated rejection (cABMR), improve renal function, reduce proteinuria, and increase graft survival without changing the immunosuppressive regimen.
  Other Names: CSM Cell Therapy
  Arms: Arm 1 (CSM Group)
Other: Placebo (NaCl 0.9%) Treatment — Patients in this arm will receive placebo treatments, which will consist of 150 mL of saline (NaCl 0.9%) administered intravenously at the same intervals as the CSM group (days 0, 7, 14, and 21). The placebo will be administered under the same conditions as the treatment, and the participants and investigators will remain blinded to the group allocation. Like the CSM group, no changes will be made to the patients' immunosuppressive regimen.
  Arms: Arm 2 (Control Group)

SUMMARY:
Kidney transplantation is the best treatment for end-stage chronic kidney disease (CKD), improving survival and quality of life, while reducing treatment costs. However, immunosuppressive therapies reduce acute rejection but have not significantly improved graft survival (60% at 10 years). Graft loss is largely due to chronic antibody-mediated rejection (cABMR), which remains a major challenge with no specific treatment. In our center, 20 cABMR cases confirmed by biopsy were identified in 2018-2019, with 40% of patients returning to dialysis.

Cellular therapies aiming at graft tolerance induction are promising strategies. The European consortium The-One-Study conducts Phase II trials using non-mesenchymal immunoregulatory cells to reduce immunosuppressive treatment and/or prevent infections or tumors. Mesenchymal Stromal Cells (MSCs), not part of this consortium, modulate the function of cells involved in acute or chronic rejection. In kidney transplantation (living donor), MSCs reduce acute rejection by 64% at 6 months, infections by 36%, with lower doses of immunosuppressants.

A recent randomized trial showed that injecting MSCs one and a half months after kidney transplantation allowed discontinuation of calcineurin inhibitors without increased rejection risk. At 6 months, there were no differences in renal function or tissue damage, indicating the potential to stop calcineurin inhibitors following MSC injection. Additionally, a significantly higher level of regulatory lymphocytes was observed. Previous attempts to discontinue calcineurin inhibitors early showed increased rejection risk.

A recent study (Neptune Phase Ib) with allogeneic MSCs demonstrated that tacrolimus doses could be reduced without acute or chronic rejection. In the cABMR model, MSC injection reduced creatinine by 45%, proteinuria by 70%, and fibrotic lesions. A study by Wei et al. showed that allogeneic bone marrow MSCs improved renal function in chronic rejection.

Given the easier availability of umbilical cord MSCs, which also have more significant paracrine activities, our goal is to demonstrate that allogeneic umbilical cord MSCs can serve as a treatment for cABMR.

DETAILED DESCRIPTION:
Currently, for patients with active chronic antibody-mediated rejection (cABMR) who do not respond to IV immunoglobulin (IV-Ig) infusions, there is no treatment that controls the rejection. Treatments targeting B lymphocytes (Rituximab) or plasma cells (Bortezomib) have not shown benefits in controlling the antibody-secreting cells and chronic rejection in most cases. A non-randomized pilot study using Tocilizumab for cABMR treatment showed a reduction in microinflammation but no modification of chronic lesions. The natural progression of the disease leads to kidney graft loss and the need for dialysis in 20-30% of transplanted patients within the first year. This technique is associated with a decrease in quality of life, frequent long-term work stoppage, increased mortality, and a rising number of patients on the waiting list, increasing the waiting time for others and the societal cost (four times higher than transplantation, about €80,000 per patient per year).

The hypothesis of this research is that Mesenchymal Stromal Cells (MSCs), with their immunomodulatory functions on all the cells involved in cABMR, may slow the progression of chronic humoral rejection that does not respond to IV-Ig. The expected benefit for patients is to gain control over chronic humoral rejection, reduce proteinuria, and extend graft function, thereby reducing the need for dialysis. Allogeneic MSCs derived from umbilical cord tissue have prolonged immunoregulatory properties and are immediately available.

Description of Knowledge Related to the Condition Kidney Transplantation and Chronic Rejection Kidney transplantation is the best treatment for chronic kidney failure, improving patient survival (about twice as long for transplant recipients compared to those on dialysis, regardless of age) and quality of life, while reducing overall treatment costs compared to hemodialysis. Dialysis costs are estimated at €80,000 per patient per year in industrialized countries, making kidney failure one of the most costly chronic diseases for society, whereas kidney transplant costs are equivalent to dialysis in the first year but become four times cheaper afterward (€20,000 per patient per year). Therefore, the additional cost of dialysis versus transplantation after the first year is €60,000 per patient per year. Currently, around 60,000 kidney transplants are performed annually worldwide, with 3,800 in France. The prevalence of patients with functioning grafts in France is around 40,000, with an average graft survival of 15 years.

It is crucial to prolong graft survival. Since the 1980s, new immunosuppressive drugs, such as anti-calcineurins, have significantly reduced the incidence of acute rejection (by 60%). The current rate of acute cellular rejection is 12-15% in the first year for non-immunized patients. However, these treatments have not significantly improved graft survival and do not prevent chronic allograft dysfunction. Thus, after the first year post-transplant, the main cause of graft loss remains chronic allograft dysfunction, occurring at a rate of 5% per year. The pathophysiology of chronic allograft dysfunction is complex, involving both immunological (acute or chronic rejection, antibody-mediated, donor-specific antibodies) and non-immunological factors (delayed graft function, infections, calcineurin toxicity, hypertension). Interstitial fibrosis and tubular atrophy are commonly observed, indicating accelerated graft aging. Significant progress has been made in characterizing the allogeneic response through improved detection techniques for alloantibodies (Luminex) and updates to the Banff classification, which is now the standard for analyzing graft histopathology.

It has been established that antibodies directed against donor HLA (Donor-Specific Antibodies, DSA) play a crucial role in both acute and chronic antibody-mediated rejection. Thus, the main cause of graft loss is chronic active antibody-mediated rejection (cABMR), and managing chronic allograft dysfunction remains one of the biggest challenges in kidney transplantation due to the lack of specific treatments. Currently, only IV-Ig infusions are used, though no definitive evidence of their effectiveness in treating acute or chronic humoral rejection has been demonstrated. Additionally, strategies targeting antibody-producing cells (memory B lymphocytes and/or plasma cells) have not proven effective due to possible escape mechanisms of these lymphocyte populations. A recent retrospective study suggested that Rituximab treatment may lead to partial improvement in a subgroup of patients with chronic humoral rejection.

Mesenchymal Stromal Cells (MSCs) Among emerging cellular therapies, Mesenchymal Stromal Cells (MSCs) are particularly promising for transplantation because of their remarkable immunosuppressive and anti-fibrotic properties. Initially described in bone marrow, MSCs can now be isolated from various tissues, including bone marrow, adipose tissue, dental pulp, and umbilical cord. MSCs derived from the Wharton's jelly of the umbilical cord (UMSCs) are particularly noted for their robust anti-inflammatory and immunomodulatory properties. These cells express mesenchymal markers such as CD73, CD90, and CD105 but do not express hematopoietic or endothelial markers, nor do they express class II HLA antigens. MSCs are multipotent and can differentiate in vitro into adipocytes, osteocytes, chondrocytes, and even myocytes and tenocytes under specific conditions. MSCs modulate the immune response by interacting with both innate and adaptive immune cells, inhibiting dendritic cell differentiation, T cell proliferation, and B cell maturation, and promoting the emergence of regulatory T cells. These effects are mediated through direct cell contact, soluble factor secretion (such as TGF-β, HLA-G, PGE2), and the synthesis of indoleamine 2,3-dioxygenase (IDO), which catabolizes tryptophan.

Given these properties, MSCs may help prevent or treat both acute and chronic rejection, and previous studies have suggested their potential in preventing acute rejection after kidney transplantation and in treating graft-versus-host disease in bone marrow transplantation.

Preclinical and Clinical Data Preclinical data have demonstrated the anti-fibrotic potential of MSCs. In 2012, the Grinyo group showed in a rat model of chronic kidney allograft rejection that MSC injection led to improved renal function, reduced proteinuria, and decreased interstitial fibrosis and tubular atrophy lesions. These results, while promising, still require further investigation to fully understand the underlying mechanisms, which are likely mediated by soluble factors. Further studies in vitro have shown that MSCs can inhibit the proliferation of renal myofibroblasts, which are key cells involved in chronic rejection. This preliminary data supports the hypothesis that MSCs could slow the progression of fibrosis in grafts during chronic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged ≥18 years
* Renal transplant recipient for ≥1 year and <10 years
* Chronic humoral rejection diagnosed by renal biopsy (Banff 2017) within the last 6 months (cpt+g score ≥ 2) with donor-specific anti-HLA antibodies (MFI<10000) and unresponsive to 3 monthly IV-IG treatments (2 g/kg) (persistence of histological lesions of Chronic Humoral Rejection; no improvement in eGFR >20%; proteinuria/creatinine ratio not regressed by more than 50% and DSA not regressed by 50%)
* eGFR (CDK-epi) > 30ml/min
* Proteinuria >1 g/24h or proteinuria/creatinine ratio >150 mg/mmol
* Patient able to attend follow-up consultations
* Patient capable of understanding and following the protocol
* Signed informed consent from the patient
* Affiliation to a social security system

Exclusion Criteria:

* Multiple transplant
* HIV-positive patient or patient with an acute or chronic uncontrolled viral infection such as hepatitis B or C
* Patient with an active bacterial infection
* Patient with decompensated heart failure or known ejection fraction <40%
* Patient with known liver cirrhosis or liver failure (Factor 5 <50%) or hepatic cytolysis (ALT >5N)
* Patient treated for a solid tumor or hematopoietic malignancy in the past 5 years, excluding skin tumors (except melanoma) (less than 3 skin tumors) BK virus nephropathy diagnosed by renal biopsy or presumed (2 BK virus PCR > 10^4 for 3 weeks) at the time of inclusion
* Pregnant woman or woman of childbearing age not using effective contraception during her participation in the study
* Patient with a known or suspected contraindication to the administration of any product used in the study, including the active substance or any excipients
* Patient deprived of liberty by judicial or administrative decision
* Adult patient under legal protection (guardianship, curatorship, or legal safeguard)
* Patient receiving psychiatric care and not stabilized
* Participation in another interventional clinical trial involving humans or in the exclusion period following a previous clinical trial involving humans (corresponding to the half-life of the experimental drug)
* Patient who received treatment with Rituximab or Velcade within the 12 months prior to inclusion and has chronic humoral rejection resistant within the past year
* Patient under state medical assistance (AME)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Umbilical Cord Allogeneic MSC Injection on Kidney Function in Patients with Chronic Active Antibody-Mediated Rejection (cABMR) | 0, 24 months
  Estimated Glomerular Filtration Rate (eGFR)

SECONDARY OUTCOMES:
Safety of MSC Injection | 0,7,14,21 day
  Oxygen saturation: Percentage (%)
Safety of MSC Injection | 0,7,14,21 day
  Dyspnea (Shortness of Breath) : Clinical assessment (scale or Yes/No)
Blood Pressure | 0,7,14,21 day
  mmHg (Systolic/Diastolic)
Estimated Glomerular Filtration Rate (eGFR) | 0,7,14,21 day
  mL/min/1.73m²
C-Reactive Protein (CRP) Levels | 0,7,14,21 day
  mg/L
Cellular Infiltration (Banff 2017 Criteria) | 0,7,14,21 day
Renal Function Evaluation | Day 0 , Month 1, Month 2, Month 6 , Month 12 , Month 18 , Month 24
  Estimated Glomerular Filtration Rate (eGFR) by CDK-EPI
Dialysis Requirement | 12 months , 24 months
  Incidence (Yes/No)
Proteinuria Evaluation | Day 0 , Month 1 , Month 2 , Month 6 , Month 12 , Month 18 , Month 24
  Grams of protein per 24 hours
Anti-HLA Antibodies Evaluation | Day 0, Month 2, Month 6, Month 12, Month 24
  Presence (Yes/No)
Renal Fibrosis Progression | 6 months
T and B Lymphocyte Phenotyping | Day 0, Month 2, Month 6
  Percentage (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Henri Mondor, Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION